CLINICAL TRIAL: NCT01051687
Title: Botulinum Toxin Treatment for Localized Vitiligo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Ghada Binsaif, King Saud University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-101
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2010-01

CONDITIONS: Vitiligo
Keywords: vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control skin patches (No Intervention): no intervention will be given to the patches
- botulinum toxin A (Active Comparator): Dilution of 1 ml of unpreserved saline per 100 U vial of BOTOX (Allergen pharmaceuticals, Irvine, CA). 2 units were injected intradermally every 1 cm2 with a 1ml syringe and 30 gauge needle.
  Interventions: Drug: Botulinum toxin A

INTERVENTIONS:
Drug: Botulinum toxin A — Dilution of 1 ml of unpreserved saline per 100 U vial of BOTOX (Allergen pharmaceuticals, Irvine, CA). 2 units were injected intradermally every 1 cm2 with a 1ml syringe and 30 gauge needle.
  For each patient with focal vitiligo, one vitiliginous patch - or two patches from different sites- will be treated. The other patches from the contra lateral site will be left untreated and used as control at the follow-up visit. For each patient with segmental vitiligo, half of the lesion will treated. The other half will be left untreated and used as a control at the follow-up visit.
  Arms: botulinum toxin A

SUMMARY:
Background: New light shed on the cholinergic aspects of vitiligo pathophysiology. It was found that acetylcholine concentration increased with a significantly reduced expression of acetylcholinesterase in vitiliginous patches that return to normal up on repigmentation.

Objective: The investigators will undertook this controlled, prospective pilot study to evaluate the efficacy and safety of botulinum toxin A in patients with localized vitiligo.

Methods: 10 patients with focal or segmental vitiligo will be recruited. For each patient with focal vitiligo, one or two vitiliginous patches will be treated. The other patches will be used as control. For each patient with segmental vitiligo, half of the lesion will be treated. The other half will be used as a control. Botulinum toxin will be injected. The response will be analyzed at the initial visit, two weeks and at two and six months after therapy.

DETAILED DESCRIPTION:
While performing a botulinum toxin A (BTX-A) treatment for glabellar frown lines and crow's feet of a lady who has also periocular vitiligo, we noted gradual and complete resolution of the vitiliginous patch, within few months, without adding other therapy. To test this observation, whether BTX-A lead to this repigmentation or it was a spontaneous one, we designed a controlled, prospective pilot study to evaluate the efficacy and safety of BTX-A in patients with localized vitiligo.

MATERIAL AND METHODS

Patients The study will be conducted in the dermatology clinic at King Khalid University Hospital. 10 patients with focal or segmental vitiligo will recruited to the study Data will be collected by patients interview included: patient characteristics (age, sex, age of onset of vitiligo, disease activity, presence of pruritus), medical history, previous treatment modalities including the clinical outcome of each modality. Complete physical examination and laboratory testing including: complete blood count, fasting blood sugar and thyroid autoantibodies were performed.

Injection Procedure Dilution of 1 ml of unpreserved saline per 100 U vial of BOTOX (Allergen pharmaceuticals, Irvine, CA). 2 units will injected intradermally every 1 cm2 with a 1ml syringe and 30 gauge needle. No other treatment modality will performed during the study.

Assessments For each patient with focal vitiligo, one vitiliginous patch - or two patches from different sites- will be treated. The other patches from the contra lateral site will be left untreated and used as control at the follow-up visit. For each patient with segmental vitiligo, half of the lesion will be treated. The other half will be left untreated and used as a control at the follow-up visit. The main outcome is the percentage of repigmentation in the previously depigmented patch, in form of color or size changes and folliculocentric repigmentation, of the treated and the control patches. Each patient will be assessed by the three investigators before and after injection with BTX-A. Patients will; be re-examined at 2 wk, 2 and 6 months after therapy. The outcome of each visit will be noted on a standardized sheet. Standardized photographs of the treated and control patches, including measurement, will be taken at each visit.

Repigmentation in previously depigmented patch will be judge by the photograph and the measurement of lesion and compared to pre treatment status by a blinded dermatologist.

ELIGIBILITY:
Inclusion Criteria:

* focal vitiligo
* segmental vitiligo

Exclusion Criteria:

* receiving any treatment during the last 4 weeks patient with contra indication to BTX-A

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
the percentage of repigmentation in the previously depigmented patch, in form of color or size changes and folliculocentric repigmentation, of the treated and the control patches. | Patients will be re-examined at 2 wk, 2 and 6 months after therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Binsaif, MD, Principal Investigator — King Saud University
Locations (1):
- King Khalid University Hospital, Riyadh, Riyadh Region, Saudi Arabia